CLINICAL TRIAL: NCT07297303
Title: Longitudinal Pulmonary Chronic Graft-versus-host-disease (GvHD) Assessment in Hematopoietic Stem Cell Transplantation (HSCT) Patients
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202501048RIND
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Bronchiolitis Obliterable Syndrome
Keywords: hematopoietic stem cell transplantation; GvHD; Obstructive airway disease; Pulmonary rehabilitation; Cardiopulmonary exercise test
MeSH Terms: conditions — Lung Diseases, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- A hematopoietic stem cell transplantation cohort

SUMMARY:
Prospective observational study on the clinical characteristics of pulmonary graft-versus-host disease in patients after hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
In patients undergoing hematopoietic stem cell transplantation (HSCT), pulmonary complications include both infectious and non-infectious conditions. Among these, bronchiolitis obliterans syndrome(BOS) represents a severe manifestation of pulmonary graft-versus-host disease. BOS typically develops within two years after HSCT, with a median time to diagnosis ranging from 6 months to 1 year. However, it may occur at any time between 50 days and 10 years post-transplantation. During the early course of the disease, many patients are asymptomatic; progressive dyspnea and cough subsequently develop, usually over weeks to months. Potential risk factors include chronic graft-versus-host disease, older age, impaired pre-transplant pulmonary function, and early respiratory infections.

The current diagnostic criteria for BOS are still based on the recommendations of the 2014 National Institutes of Health Consensus on chronic graft-versus-host disease. Treatment for BOS remains complex and is supported by limited evidence. In Taiwan, local data on pulmonary complications-particularly BOS-remain insufficient.

We aim to establish a prospective cohort study enrolling approximately 600 participants to analyze the epidemiology, clinical manifestations, pulmonary function changes (including impulse oscillometry), imaging findings, and biomarker alterations associated with pulmonary graft-versus-host disease in Taiwanese HSCT recipients.

ELIGIBILITY:
Inclusion Criteria:

1. Age>18
2. Will Receive first time Allo-HSCT patients

Exclusion Criteria:

1. Respiratory failure
2. Hemodynamic unstable
3. Pneumothorax or bronchial fistula
4. Acute coronary syndrome in recent 1 month
5. The patient couldn't walk longer than 20 m
6. Severe lower-limb arthropathy
7. The patient couldn't cooperate well
8. Need all-day oxygen supplement
9. The patient received lung transplantation before

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At National Taiwan University Hospital and National Taiwan University Hospital Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of bronchiolitis obliterans syndrome | From enrollment to the end of treatment at 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to privacy concerns and limitations specified by the ethics committee/institutional review board.